CLINICAL TRIAL: NCT03997279
Title: Double-blind, Placebo-controlled, Randomized Study for Assesment of the Efficiency and Safety Quadruple Therapy for Helicobacter Pylori Infection With or Without the Addition of Saccharomyces Boulardi Probiotic
Brief Title: Assesment of the Efficiency and Safety Helicobacter Pylori Therapy With or Without Saccharomyces Boulardii
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Miodrag Krstic, Clinical Professor, Clinical Centre of Serbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AB-2019-4
Record Dates: First submitted 2019-06-12; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; Saccharomyces boulardi; Eradication therapy
MeSH Terms: interventions — Rabeprazole; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S.boulardi (Experimental): Quadruple eradication therapy with S. boulardi
  Interventions: Drug: Saccharomyces boulardii
- Placebo (Placebo Comparator): Quadruple eradication therapy without S. boulardi
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saccharomyces boulardii — Rabeprazole 20 mg 2x1, for 14 days, followed by 1x1 for 14 days, Amoxicillin 1000 mg 2x1, for 14 days, Clarithromycin 500 mg 2x1, for 14 days, Metronidazole 500 mg 2x1, for 14 days, Saccharomyces boulardi 500 mg 1x1, for 3 week
  Other Names: Rabeprazole; Amoxicillin; Clarithromycin; Metronidazole
  Arms: S.boulardi
Drug: Placebo — Rabeprazole 20 mg 2x1, for 14 days, followed by 1x1 for 14 days, Amoxicillin 1000 mg 2x1, for 14 days, Clarithromycin 500 mg 2x1, for 14 days, Metronidazole 500 mg 2x1, for 14 days, Placebo 1x1, for 3 week
  Other Names: Rabeprazole; Amoxicillin; Clarithromycin; Metronidazole
  Arms: Placebo

SUMMARY:
This study assesses the effect of quadruple therapy for H. pylori, with the addition of probiotics Saccharomyces boulardii. In addition, he assesses whether this combination reduces the frequency of adverse effects of eradication therapy, and whether it affects the compliance.

DETAILED DESCRIPTION:
Standard triple therapy for H. pylori infection proved to be insufficiently effective, primarily due to antibiotics resistance.Therefore, the latest Maastricht consensus suggests using bismuth-quadruple or non-bismuth-quadruple therapy, in regions with high clarithromycin resistance. The addition of probiotics with eradication therapy has never become a standard treatment. However, the Maastricht consensus suggest that the addition of probiotics could increase the effectiveness of quadruple therapy.

The study was designed as a prospective, double-blind, randomized, case-control intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Dyspepsia
* Patients not treated for H. Pylori
* Age of 18-50 years
* Positive urea breath test

Exclusion Criteria:

* Alarm symptoms (anemia, persistent vomiting, hematemesis, dysphagia, significant weight loss, palpable mass in abdomen)
* Gastric cancer
* Immunosuppressive therapy
* Use of acetylsalicylic acid
* Severe renal failure
* Severe liver failure
* Immunodeficiency
* Proven malignant disease
* Penicillin allergy
* Allergy to any component of dietary supplement (Saccharomyces boulardii and Vitamin D)
* Chronic alcoholism
* Pregnancy
* Lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Result of urea breath test (Eradication of H.pylori) | baseline to 8 weeks after the introduction of the therapy
  Test remains positive (Eradication of H.pylori unsuccessful) or test becomes negative (eradication of H.pylori successful)

SECONDARY OUTCOMES:
Side effects of eradication therapy | baseline to 8 weeks after the introduction of the therapy
  Number and severity of adverse events of standard eradication therapy
Compliance of eradication therapy | baseline to 8 weeks after the introduction of the therapy
  Patient successfully completed prescribed therapy